CLINICAL TRIAL: NCT00861718
Title: A Phase I, Single-center, Double-blind, Randomized, Placebo-controlled Study to Assess the Safety, Tolerability, and Pharmacokinetics of AZD7268 When Given in Multiple Ascending Oral Doses in Healthy Subjects
Brief Title: Phase I Multiple Ascending Dose Study for AZD 7268 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Mark A. Smith, M.D., AstraZeneca Pharmaceuticals
Allocation: Randomized | Model: Single Group | Masking: Quadruple
Other Study IDs: D1151C00003
Record Dates: First submitted 2009-03-12; First posted 2009-03-13 (Estimated); Last update posted 2009-12-10 (Estimated); Status verified 2009-12

CONDITIONS: Healthy
Keywords: Phase 1; Healthy Volunteer

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- AZD7268 (Experimental)
  Interventions: Drug: AZD7268
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD7268 — Capsule, Oral, QD
  Arms: AZD7268
Drug: AZD7268 — Capsule, Oral, BID
  Arms: AZD7268
Drug: Placebo — Capsule, Oral BID
  Arms: Placebo

SUMMARY:
Multiple Ascending Dose Study

ELIGIBILITY:
Inclusion Criteria:

* Provision of Informed Consent
* Healthy male subjects and female subjects (of non-child bearing potential)

  * with suitable veins for cannulation or repeated venipuncture

Exclusion Criteria:

* Inability to understand or cooperate with given information
* Any positive result on screening for human immune deficiency virus (HIV), Hepatitis B, or Hepatitis C test
* History of seizure (including infancy febrile seizures) or family history of seizure

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2009-04; Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
To assess the safety and tolerability of AZD7268 when given orally in multiple ascending doses to healthy male subjects and female subjects of non-childbearing potential. | Safety assessments are made at each visit, at least daily, during the study.

SECONDARY OUTCOMES:
To characterize the pharmacokinetics of AZD7268 in plasma. | Serial blood samples for pharmacokinetic analysis will be collected on Days 1,2,3 and Days 9, 10, and 11 of the study. Additional pharmacokinetic samples will be collected on Days 6, 7, and 8

CONTACTS AND LOCATIONS:
Overall Officials: Sylvan Hurewitz, M.D., Principal Investigator — AstraZeneca Clinical Pharmacology Unit, US
Locations (1):
- Research Site, Philadelphia, Pennsylvania, United States